CLINICAL TRIAL: NCT03799458
Title: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) for Sensory Deficits in Complex Traumatic Brain Injury
Acronym: NAVIGATE-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Biomedical Research Institute of New Mexico (Other); New Jersey Institute of Technology (Other); University of Miami (Other); The Mind Research Network (Other); The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDMRP-PT160096
Record Dates: First submitted 2018-12-12; First posted 2019-01-10 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: 120 subjects will be recruited for this study: 40 healthy controls subjects for the imaging-only group, and 80 mTBI subjects for the stimulation arm who have suffered mild TBI at least 3 months prior to study enrollment, but not more than 15 years prior to enrollment. The 80 mTBI subjects will be randomized to either active stimulation (40) or sham stimulation (40).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Active and sham HD-tDCS will be delivered with the same device, and participants and research technician are blinded to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Active Stimulation (Active Comparator): Active HD-tDCS will be delivered while subjects perform sensory training tasks.
  Interventions: Device: Active High-definition transcranial direct current stimulation (HD-tDCS)
- Sham Stimulation (Sham Comparator): Sham HD-tDCS will be delivered while subjects perform sensory training tasks.
  Interventions: Device: Sham High-definition transcranial direct current stimulation (HD-tDCS)
- Imaging Only (No Intervention): 40 subjects will undergo initial testing only as a healthy control group.

INTERVENTIONS:
Device: Active High-definition transcranial direct current stimulation (HD-tDCS) — Active HD-tDCS delivers active current through 2-10 electrodes held against the scalp with a lycra cap at specified 10-20 electroencephalography (EEG) coordinates.
  Arms: Active Stimulation
Device: Sham High-definition transcranial direct current stimulation (HD-tDCS) — Sham HD-tDCS delivers sham current through 2-10 electrodes held against the scalp with a lycra cap at specified 10-20 electroencephalography (EEG) coordinates
  Arms: Sham Stimulation

SUMMARY:
Aim 1: To use magnetoencephalography (MEG) and magnetic resonance imaging (MRI) in Veterans and civilians with mild traumatic brain injury (mTBI) and sensory postconcussive symptoms (PCS) to demonstrate the mechanism of therapeutic benefit of HD-tDCS for sensory symptoms, as shown by reliable changes in the activity of the cognitive control network (CCN) and sensory system network (SSN) following stimulation; Aim 2: this intervention will result in long-term improvements in measures of executive function, depression/anxiety, and quality of life.

DETAILED DESCRIPTION:
Experimental Design and Methods Participants: 120 subjects will be recruited for this study from the NM VA Health Care System and community, 40 healthy controls subjects for an imaging-only group, and 80 mTBI subjects for the stimulation arm who have suffered injury at least 3 months prior to study enrollment, but not more than 15 years prior to enrollment. All participants will be 18-59 years of age.

Recruitment: Human participants (ages 18-59) will be invited to come to the University of New Mexico (UNM) to ask questions prior to providing consent. They will be provided with consent forms that describe the study procedures and potential risks.

Once informed consent is obtained and the appropriate forms signed, the participant will be assigned a unique research subject identifier (URSI) number, and from that point forward all research data will only be labeled with the URSI number. The key linking identifiers of participants to the URSI will be maintained on a separate database that will be stored behind locked doors, in a locked filing cabinet in a secure area. All participants may then undergo demographic data collection, neuropsychological assessments sensory evaluation, at UNM. They may also undergo MEG and MRI at the Mind Research Network (MRN), located in the same building.

Demographic Data: As part of the initial assessment, basic demographic data regarding the subject may be noted down, including age, gender, socioeconomic status, educational attainment, handedness, use of common stimulants such as caffeine, and brain injury severity. They may also be asked if they are willing to allow their medical record to be accessed, for the purposes of confirming details about any traumatic brain injury (TBI) as well as obtaining results of neuroimaging studies done at the time of injury or afterward. This will include medical, surgical, neurological and psychiatric history, results of lab tests, brain scans, electroencephalography tests, medication lists, information from doctor's visits and hospital visits.

Neuropsychological testing procedures: All neuropsychological testing will be administered in the Center for Brain Recovery and Repair Core by trained study personnel under direct supervision of core directors. The following domains and tests will be administered: Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (Examiner); Digit Span; Delis-Kaplan Executive Function Systems (DKEFS) Trail-making Test Conditions 2 and 4; Hopkins Verbal Learning Test (HVLT); Frontal Systems Behavior Scale (FrSBe); Test of Memory Malingering (TOMM); Wechsler Test of Adult Reading (WTAR); Digit Symbol Coding; Handedness; Socioeconomic Status (SES); Patient's Global Impression of Change (PGIC); Glasgow Outcome Scale-Extended (GOSE).

Sensory Assessment: Hearing, balance, and vision will be assessed using Common Data Element (CDE) instruments, including the Hearing Handicap Assessment, the Test for Visual Discomfort, the modified Balance Error Scoring System. Oculomotor control will be assessed using virtual reality goggles (Oculus) with implanted eye trackers (iScan).

Magnetoencephalography: Magnetoencephalography (MEG) may be done after neuropsychological testing. The participant will sit in the MEG scanner to record brain magnetic fields. MEG setup takes between 10 and 30 minutes, and subsequent recording takes one hour. During MEG assessments participants will complete numerous tasks. Each task is designed to parse different cognitive mechanisms that contribute to sensory performance. In perceptual tasks, participants will discriminate tone pitches amongst novel distracting tones (Auditory Orienting Task; AOT). For eye movement tasks, participants are asked look either towards or away from a visual stimulus (Pro- and Anti-saccades).

Magnetic resonance imaging (MRI): MRI scan(s) will be obtained for integration with MEG, as needed for analyses. Total scan time, including participant setup and removal, is expected to take 1 hour. Participants may lie down on a table and be placed into a long donut-shaped magnet. During the scan, participants will be asked to rest quietly or to fixate on a dot on a screen in front of them, or to perform a memory task. No contrast will be used. Any female over 18 who thinks she may be pregnant will complete a urine pregnancy screen before the MRI scan.

Following initial testing, the participants in the stimulation arm of the study will receive 10 consecutive weekday sessions of high-definition transcranial direct current stimulation. 2 milliamperes active or sham anodal current will be delivered to the left dorsolateral prefrontal cortex for 30 minutes. During this time, participants will perform vision therapy tasks through a virtual reality headset, or a computer-based working memory task. Skin sensations will be assessed every 10 minutes.

Post stimulation testing: the next available weekday following completion of the study protocol, subjects will return to UNM to repeat the demographic, neuropsychological, sensory, and imaging assessments.

Long term followup: At 1 month, 3 months and 6 months after stimulation, subjects will be contacted via telephone or meet in person, and will be administered the Beck Depression Inventory (BDI-II), Posttraumatic Stress Disorder Checklist-Military (PCL-M), the Neurobehavioral Symptom Inventory (NSI), and Patient Global Impression of Change (PGIC) quality of life assessment tools utilized before and immediately after, after stimulation. Veterans will undergo these study followup visits at NMVAHCS, and civilians at UNM.

ELIGIBILITY:
Inclusion Criteria:

1. are US Veteran or Active Duty Military personnel aged 18-59,
2. have suffered a mild TBI (alteration in neurological functioning < 24 hours, loss of consciousness (LOC) less than 30 minutes, Glasgow coma scale (GCS) score (if available) of between 13 and 15 acutely, and less than 24 hours of post-traumatic amnesia (PTA));
3. were injured between 3 months and 15 years ago;
4. have post-traumatic sensory symptoms as evidenced by endorsing at least 2 out of 12 sensory symptoms on the Neurobehavioral Symptom Inventory (NSI), a measure of post-traumatic symptoms from the NIH Common Data Elements (CDE) to a severity of "3" or higher,
5. are fluent in English,
6. have been on stable doses of any psychotropic medications for the past 2 months.
7. The imaging-only group will have the same inclusion and exclusion criteria except they will not have had a head injury.

Exclusion Criteria:

1. any history of moderate or severe TBI;
2. a prior history of other neurological disease or any history of seizures beyond immediate post-traumatic seizure, to as to reduce risk of exacerbation of epilepsy or other neurological symptoms;
3. history of psychosis, so as to reduce risk of psychiatric decompensation;
4. history of current or recent (within two years) substance/alcohol dependence, to reduce confounding effects on cognition and plasticity;
5. any discontinuity in skull electrical conductivity (i.e., unhealed burr holes in scalp) or artificially constructed (metal or plastic) craniotomy cover, to reduce risk of unimpeded electrical current;
6. presence of any implanted electrical device (e.g. pacemaker), to reduce risk of device malfunction;
7. recent medical hospitalization (within three weeks), to reduce risk of medical decompensation during the study;
8. any condition that would prevent the subject from completing the protocol; 9) appointment of a legal representative, as assessed via direct inquiry of the subject and a designated trusted other, to avoid coercion of a vulnerable population;

10) any significant blindness, to screen out peripheral sensory damage; 11) any significant deafness beyond mild hearing loss, to screen out peripheral sensory damage; 12) any ongoing litigation related to TBI, to prevent interference with legal proceedings; 13) any contraindication to MRI; 14) membership in an identified vulnerable population, including minors, pregnant women, and prisoners, so as to prevent coercion.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, including demographic, neuropsychological, and imaging data, will be uploaded to FITBIR for use by TBI researchers, as specified by the grant sponsor.
Time Frame: Data will be uploaded to the Federal Interagency Traumatic Brain Injury Registry (FITBIR) at study termination.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Stimulation | Sham Stimulation | Imaging Only
Started | 21 | 21 | 37
Completed | 11 | 10 | 29
Not Completed | 10 | 11 | 8

BASELINE CHARACTERISTICS:
Population: This is the population of patients with complete behavioral and magnetoencephalography data
Groups:
- Active Stimulation TBI Group: Subjects have experienced a mild TBI with ongoing symptoms. Active HD-tDCS will be delivered while subjects perform sensory training tasks.
  Active HD-tDCS delivers active current through 2-10 electrodes held against the scalp with a lycra cap at specified 10-20 electroencephalography (EEG) coordinates. Sham delivers a negligible amount of current that does not cause physiological changes.
- Sham Stimulation TBI Group: Subjects have experienced a mild TBI with ongoing symptoms. Sham HD-tDCS will be delivered while subjects perform sensory training tasks.
  Active HD-tDCS delivers active current through 2-10 electrodes held against the scalp with a lycra cap at specified 10-20 electroencephalography (EEG) coordinates. Sham delivers a negligible amount of current that does not cause physiological changes.
- Imaging Only Control Group: Subjects will undergo initial testing only as a healthy control group.
- Total: Total of all reporting groups
Arm/Group | Active Stimulation TBI Group | Sham Stimulation TBI Group | Imaging Only Control Group | Total
Number analyzed (Participants) | 11 | 10 | 28 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (10.1) | 49.7 (10.5) | 51.4 (13.2) | 49.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 11 | 13
  Male | 10 | 9 | 17 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 10 | 18
  Not Hispanic or Latino | 8 | 5 | 18 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 7 | 18 | 35
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 28 | 49
Neurobehavioral Symptom Inventory Somatic Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The NSI is a validated scale of postconcussive symptoms; the Somatic Subscale score captures severity of physical symptoms such as tinnitus, blurry vision, loss of balance, and insomnia. (range 0-48; 0-12 mild; 13-24 moderate; 25-36 severe; 37-48 very severe)
  units on a scale | 19.9 (10.5) | 18.9 (11.3) | 2.9 (3.3) | 10.0 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Postconcussive Sensory Symptoms
Description: The NSI is a validated scale of postconcussive symptoms; the Somatic Subscale score captures severity of physical symptoms such as tinnitus, blurry vision, loss of balance, and insomnia. (range 0-48; 0-12 mild; 13-24 moderate; 25-36 severe; 37-48 very severe)
Time Frame: 2 week visit
Population: For active and sham, analysis population includes all participants who completed intervention and all pre-intervention and post-intervention visit assessments. For imaging only group, analysis includes all participants who completed all pre-intervention visit assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation | Imaging Only
Number analyzed (Participants) | 11 | 10 | 28
score on a scale
  Pre-Intervention (baseline visit) | 19.9 (10.5) | 18.9 (11.3) | 2.9 (3.3)
  Post-Intervention (2 week visit): number analyzed (Participants) | 11 | 10 | 0
  Post-Intervention (2 week visit) | 20.6 (9.4) | 17.5 (9.5) |

2. Secondary Outcome: Magnetoencephalography Peak Activation
Description: Peak activation during the Auditory Orienting Task (AOT) performed during magnetoencephalography
Time Frame: 2 week visit
Population: For active and sham intervention groups, analysis population includes all participants who completed intervention
Measure: Mean (Standard Deviation); unit: femtotesla
Arm/Group | Active Stimulation | Sham Stimulation | Imaging Only
Number analyzed (Participants) | 11 | 10 | 28
femtotesla
  Pre-Intervention (baseline visit) | 3.07 (0.87) | 3.49 (0.92) | 3.31 (0.90)
  Post-Intervention (2 week visit): number analyzed (Participants) | 11 | 10 | 0
  Post-Intervention (2 week visit) | 3.68 (1.42) | 3.46 (1.03) |

ADVERSE EVENTS:
Time Frame: adverse event data was collected for the "Active Stimulation" and "Sham Stimulation" Arms during the 2-week stimulation period between Visit 1 and Visit 2; adverse event data were collected over a single day at Baseline for participants in the "Imaging Only" Arm.
Arm/Group | Active Stimulation | Sham Stimulation | Imaging Only
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/37
Other Adverse Events (participants affected / at risk) | 3/21 | 2/21 | 0/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (N=21) | Sham Stimulation (N=21) | Imaging Only (N=37)
syncope (Nervous system disorders) | 1 (1) | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0
headache (Nervous system disorders) | 1 (1) | 1 (1) | 0
nightmares (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03799458/Prot_SAP_000.pdf